CLINICAL TRIAL: NCT05130372
Title: Comparison of The Acute Effects of Different Stretching Techniques on Ankle Joint Range of Motion In Healthy Older Adults: A Randomised Controlled Trial
Brief Title: Comparison of The Acute Effects of Different Stretching Methods on Ankle Joint Range In Healty Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Nursen İlçin (Unknown); Ceren Devrim Şahin (Unknown)
Responsible Party: Principal Investigator, Kutay Kaslı, Kutay Kaşlı, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/17-39
Record Dates: First submitted 2021-11-08; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Older Adults; Range of Motion; Ankle Injuries
Keywords: older adults; ankle joint range of motion; roller massage; static stretching; PNF stretching
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Arm 1:Static Stretching Group Arm 2: PNF Stretching Method Group Arm 3:Roller Massager Group
Who Masked: Investigator, Outcomes Assessor
Masking Description: A single-blind, assessor-blinded, randomized controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static Stretching Group (Active Comparator): The static stretching method was actively applied while standing.The person was positioned facing the wall, supporting the wall with both hands, with the dominant foot behind. The point where a feeling of tension in the plantar flexor muscles was created and held in this position for 30 seconds. Afterward, a 15-second rest break was given. After completing 3 repetitions (3x30sec) in total, measurements were started.
  Interventions: Other: Static Stretching Method Group
- PNF Stretching Method Group (Active Comparator): The person was positioned supine, and the ankle joint was dorsiflexed by the physiotherapist to the point where the tension was felt. Then, while the person was trying to push the foot towards the plantarflexion direction for 10 seconds, the movement was prevented by the physiotherapist and isometric contraction was achieved at 20% of the maximum voluntary contraction. After 10 seconds, the person was asked to relax slowly and passive stretching was applied to the plantar flexors for 20 seconds. The contract-relax technique was applied for 30 seconds and completed with 3 repetitions (3x30sec) with 15-second rest intervals.
  Interventions: Other: PNF Stretching Method Group
- Myofascial Relaxation Method Group (Active Comparator): A comfortable position was achieved by placing a rolled towel on the front of the ankle. The roller was massaged along with the plantar flexors for 30 seconds. The movement of the cylinder from bottom to top and from top to bottom was done for a second. Three repetitions were completed (3x30sec) with a 15-second rest break. For the pressure of the roller to be stable during the application, the numbered pain scale was shown to the participants, and attention was paid to ensure that the perceived severity was 7/10 according to the numbered pain scale. Participants with dry skin in the application area were asked to moisturize with cream beforehand to avoid complications.
  Interventions: Other: Myofascial Relaxation Method Group- Roller Massage

INTERVENTIONS:
Other: Static Stretching Method Group — Static stretching has been the most common stretching method applied to the ankle in healthy older adults, and different protocols have proven to increase ankle range of motion. In this study, the static stretching method was actively applied while standing.
  Arms: Static Stretching Group
Other: PNF Stretching Method Group — The contract-relax technique was used in the PNF stretching method.
  Arms: PNF Stretching Method Group
Other: Myofascial Relaxation Method Group- Roller Massage — A theraband roller massager (Theraband®, The Hygenic Corporation, Akron, OH) was used for the myofascial relaxation method.
  Arms: Myofascial Relaxation Method Group

SUMMARY:
Introduction: To compare the acute effects of different stretching methods on ankle joint range of motion (ROM) in older adults.

Methods: A total of 78 subjects aged 65 years and older were randomly divided into three groups. After the 5-minute walk, the randomly assigned method was applied. Static Stretching Group; static stretching in 3x30sec, PNF Stretching Group; PNF contract-relax in 3x30sec and Roller Massage Group; roller massage in 3x30sec was performed. Immediately after the application, 10 minutes and 20 minutes after application, the range of motion of the ankle joint was measured in the weight-bearing lunge position.

DETAILED DESCRIPTION:
It is planned to single-blind, randomized controlled study with before-after measurements. Considering the acute effects of stretching exercise for ankle dorsiflexion in older women, the effect size was calculated as 1.02. According to this effect size, it was planned to recruit 26 people to each group with 95% confidence level and 95% power, and 78 people in total would participate in the study. Ethics committee approval of the study was received from Dokuz Eylul University Non-Interventional Research Ethics Committee (with the decision number 2017/17-39 in the meeting dated 22.06.2017). The study was conducted under the Declaration of Helsinki standards. The participants were informed about the study by the physiotherapist and all the participants provided written informed consent to participate in the study. The study included healthy and voluntary older adults aged 65 and over who were able to walk without using an assistive device, independent in their daily life activities, and scored 23 and above according to the mini-mental state test in the study. The exclusion criteria of the study were the presence of a neurological, orthopedic or cardiovascular disease affecting the lower extremity, pain or limitation of movement in the ankle joint, skin diseases, history of falling in the last 1 year, any problem that may prevent lying prone and participation in a regular exercise program. Individuals meeting the inclusion criteria were randomly assigned to one of two different groups with the help of the Random Numbers Table. The study was terminated when the target number of participants (n=78) was reached. Static stretching was applied to the first group (n=26), PNF stretching to the second group (n=26), and roller massage to the third group (n=26). Individuals meeting the inclusion criteria were randomly assigned to one of two different groups with the help of the Random Numbers Table. The study was terminated when the target number of participants (n=78) was reached. Static stretching was applied to the first group (n=26), PNF stretching to the second group (n=26), and roller massage to the third group (n=26). (Figure 1) After the stretching method to be applied was determined randomly, the participants were asked to walk for 5 minutes in a 50-meter corridor. After warming up with this light-paced walking, applied one of the three methods. Immediately after the application, 10 minutes and 20 minutes after application, the range of motion of the ankle joint was measured in the weight-bearing lunge position.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and voluntary older adults aged 65 and over
* Who were able to walk without using an assistive device,
* Independent in their daily life activities
* Who scored 23 and above according to the mini-mental state test.

Exclusion Criteria:

* Presence of a neurological, orthopedic or cardiovascular disease affecting the lower extremity,
* Pain or limitation of movement in the ankle joint,
* Skin diseases,
* History of falling in the last 1 year,
* Any problem that may prevent lying prone
* participation in a regular exercise program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Range of motion | Baseline
  The ankle ROM measurement made in the standing load-bearing position and the measurement made in the weight-bearing position.
Range of motion | Immediately after application
  The ankle ROM measurement made in the standing load-bearing position and the measurement made in the weight-bearing position.
Range of motion | 10 minutes after application
  The ankle ROM measurement made in the standing load-bearing position and the measurement made in the weight-bearing position.
Range of motion | 20 minutes after application
  The ankle ROM measurement made in the standing load-bearing position and the measurement made in the weight-bearing position.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Devrim Şahin, MSc, Study Director — Dokuz Eylul University; Nursen İlçin, Assoc. prof., Study Chair — Dokuz Eylul University; Kutay Kaşlı, MSc, Principal Investigator — Çankırı Karatekin University
Locations (2):
- Turkey (Türkiye) (2):
  - Izmir Provincial Health Directorate State Hospital, Izmir, Urla
  - Izmir Provincial Health Directorate Urla State Hospital, Izmir, Urla

IPD SHARING:
Plan to Share IPD: Undecided
It will be shared if it is in line with the objectives of the study.